CLINICAL TRIAL: NCT06269523
Title: Effects of Rehabilitation and Kinesio Taping to Prevent Axillary Web Syndrome After Breast Cancer Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Palermo (Other)
Responsible Party: Principal Investigator, Prof.ssa Giulia Letizia Mauro, Professor, University of Palermo
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: MFR032024
Record Dates: First submitted 2024-02-01; First posted 2024-02-21 (Actual); Last update posted 2024-02-21 (Actual); Status verified 2023-11

CONDITIONS: Axillary Web Syndrome
Keywords: Axillary Web Syndrome; Kinesio taping; Lymphatic drainage; Breast cancer surgery; Proprioceptive re-education
MeSH Terms: interventions — Manual Lymphatic Drainage

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment group (Active Comparator): 18 sessions of functional and proprioceptive re-education, manual lymphatic drainage associated with kinesio taping.
  Interventions: Other: Kinesio taping, Lymphatic drainage
- Control group (Active Comparator): 18 sessions of functional and proprioceptive re-education and manual lymphatic drainage.
  Interventions: Other: Lymphatic drainage

INTERVENTIONS:
Other: Kinesio taping, Lymphatic drainage — Kinesio tape, is an elastic cotton strip with an acrylic adhesive that is purported to ease pain and disability from athletic injuries and a variety of other physical disorders. The application of Kinesio Tex Tape facilitates the opening of microvalves due to a dynamic pressure variation due to alteration in skin density. This decompression activates lymphatics in the dermis and improves lymphatic flow. The end result is a tissue inflammation and swelling reduction.It has been applied at the end over every session after lymphatic dreinage (see below).
  Arms: Treatment group
Other: Lymphatic drainage — Lymphatic drainage is a type of manual manipulation of the skin based on the hypothesis that it will encourage the natural drainage of the lymph, which carries waste products away from the tissues back toward the heart. The lymph system depends on intrinsic contractions of the smooth muscle cells in the walls of lymph vessels (peristalsis) and the movement of skeletal muscles to propel lymph through the vessels to lymph nodes and then to the lymph ducts, which return lymph to the cardiovascular system. Manual lymph drainage uses a specific amount of pressure and rhythmic circular movements to stimulate lymph flow.
  Arms: Control group

SUMMARY:
Axillary web syndrome (AWS) is a complication associated with breast cancer surgery, characterized by pain, functional limitation of the shoulder and decreased quality of life. There are several physical treatment options to reduce pain and improve the functionality of the upper limb in women with AWS. This study evaluates the effectiveness of an early rehabilitation approach to prevent axillary web syndrome consisting in functional and proprioceptive re-education, manual lymphatic drainage and kinesio taping after breast cancer surgery.

DETAILED DESCRIPTION:
Axillary web syndrome (AWS), is a complication associated with breast cancer surgery, characterized by pain, functional limitation of the shoulder and decreased quality of life. The pain is localized in the axillary area and along the arm, with the limitation of the glenohumeral joint (GO) and the presence of one or more "cords" of tissue visible or palpable with the abduction of the GO, at the level of the axilla , which can extend medially up to the wrist. Incidence, etiopathogenesis and ideal treatment of this condition are not yet clear.

The literature provides several physical treatment options for AWS. Physical therapy is effective in reducing pain and improving the functionality of the upper limb. Manual lymphatic drainage is indicated in forms of lymphedema due to axillary lymphadenectomy. The commonly used rehabilitation treatment consists of functional re-education of the shoulder, neuromotor and proprioceptive re-education of the upper limb, lymphatic drainage. Kinesio taping is rarely used and not in association with rehabilitation. This study evaluates the effectiveness of an early rehabilitation approach consisting of functional and proprioceptive re-education, manual lymphatic drainage and kinesio taping after quadrantectomy and lymphadenectoma surgery for breast cancer in the prevention of axillary web syndrome.

At the U.O.C. of Functional Recovery and Rehabilitation Department of the Paolo Giaccone University Hospital in Palermo, have been enrolled 18 women between the ages of 45 and 65 years old with a diagnosis of breast cancer, underwent to quadrantectomy and axillary lymphadenectomy.

Patients have been randomly divided into two groups: treatment group, in which kinesio taping has been applied, associated with a rehabilitation protocol lasting 18 sessions of functional and proprioceptive re-education and manual lymphatic drainage; control group, subjected to 18 sessions of functional and proprioceptive re-education, manual lymphatic drainage.

Patients have been evaluated: one week after surgery (T0), at the end of the 18 sessions (T1) and 3 months after surgery (T2).

The investigators evaluated: joint excursion shoulder's degree by a goniometer; the pain, using NRS scale; muscular strength of the upper limbs using a dynamometer (PINCH GAUGE); upper limbs circumference (cyrtometry) by a meter; and the functional capacity of the shoulder, using the Constant Murley scale.

ELIGIBILITY:
Inclusion Criteria:

* women between the ages of 45 and 65 years with diagnosis of breast cancer underwent to quadrantectomy and axillary lymphadenectomy.

Exclusion Criteria:

* metastatic disease, infections, past TVP, embolia.

Ages: 45 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2021-07-21 (Actual); Primary Completion 2023-01-31 (Actual); Study Completion 2024-01-31 (Actual)

PRIMARY OUTCOMES:
NRS Scale | one week after surgery(T0)- 5 weeks after surgery(T1)-12 weeks after surgery (t2)
  NRS scale is an 11-point unidimensional scale that evaluates the intensity of pain in adults.The scale is composed of a horizontal line, with an interval ranging from 0 to 10, corresponding respectively to "no pain" and "worst pain imaginable".
Joint excursion shoulder | one week after surgery(T0)-5 weeks after surgery(T1)- 12 weeks after surgery (t2)
  Range of motion of the shoulder taken with the use of a goniometer
Muscular strength of the upper limbs | one week after surgery(T0)- 5 weeks after surgery(T1) -12 weeks after surgery (t2)
  Distal strength can be semiquantitatively measured with a dynamometer. Dynamometry is a more precise measurement of the force that a muscle can exert and can allow for differences in strength to be recorded over time.

SECONDARY OUTCOMES:
Constant Murley Score | one week after surgery(T0)- 5 weeks after surgery(T1)-12 weeks after surgery(t2)
  The Constant-Murley score (CMS) is a 100-points scale composed of a number of individual parameters. These parameters define the level of pain and the ability to carry out the normal daily activities of the patient.The Constant-Murley score was introduced to determine the functionality after the treatment of a shoulder injury. The test is divided into four subscales: pain (15 points), activities of daily living (20 points), strength (25 points) and range of motion: forward elevation, external rotation, abduction and internal rotation of the shoulder (40 points).The higher the score, the higher the quality of the function.
upper limbs circumferenze (cyrtometry) | one week after surgery(T0)- 5 weeks after surgery(T1)- 12 weeks after surgery (t2)
  measurement of the circumference of the upper limb in some points(metacarpophalangeal joint, wrist, elbow, -14 cm from the lateral epicondyle of the elbow, -7 cm from the lateral epicondyle of the elbow), elbow (+7 cm from the lateral epicondyle, +14 cm from the lateral epicondyle) with a measuring tape in centimeters.

CONTACTS AND LOCATIONS:
Locations (1):
- Functional Recovery and Rehabilitation Unit of the A.O.U.P. Paolo Giaccone, Palermo, Italy

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code

REFERENCES:
- [Background] Moskovitz AH, Anderson BO, Yeung RS, Byrd DR, Lawton TJ, Moe RE. Axillary web syndrome after axillary dissection. Am J Surg. 2001 May;181(5):434-9. doi: 10.1016/s0002-9610(01)00602-x. PMID 11448437
- [Background] Agostini F, Attanasi C, Bernetti A, Mangone M, Paoloni M, Del Monte E, Mammucari M, Maggiori E, Russo D, Marzo RD, Migliore A, Paolucci T. Web Axillary Pain Syndrome-Literature Evidence and Novel Rehabilitative Suggestions: A Narrative Review. Int J Environ Res Public Health. 2021 Oct 2;18(19):10383. doi: 10.3390/ijerph181910383. PMID 34639683
- [Background] Dinas K, Kalder M, Zepiridis L, Mavromatidis G, Pratilas G. Axillary web syndrome: Incidence, pathogenesis, and management. Curr Probl Cancer. 2019 Dec;43(6):100470. doi: 10.1016/j.currproblcancer.2019.02.002. Epub 2019 Mar 15. PMID 30898366
- [Background] Ezzo J, Manheimer E, McNeely ML, Howell DM, Weiss R, Johansson KI, Bao T, Bily L, Tuppo CM, Williams AF, Karadibak D. Manual lymphatic drainage for lymphedema following breast cancer treatment. Cochrane Database Syst Rev. 2015 May 21;2015(5):CD003475. doi: 10.1002/14651858.CD003475.pub2. PMID 25994425
- [Background] Kasawara KT, Mapa JMR, Ferreira V, Added MAN, Shiwa SR, Carvas N Jr, Batista PA. Effects of Kinesio Taping on breast cancer-related lymphedema: A meta-analysis in clinical trials. Physiother Theory Pract. 2018 May;34(5):337-345. doi: 10.1080/09593985.2017.1419522. Epub 2018 Jan 8. PMID 29308967